CLINICAL TRIAL: NCT00572299
Title: Glucocorticoids Promote Osteoclast Survival
Status: Terminated | Type: Observational
Why Stopped: Terminated due to recruitment problems
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 28727; VA Merit Review Grant (Other Grant/Funding Number: VA Merit Grant Review)
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Osteoporosis
Keywords: glucocorticoids, prednisone, alendronate,osteoclasts
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate; Prednisone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bone biopsy specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- glucocorticoids: patients receiving glucocorticoid treatment
- glucocorticoids and bisphosphonates: patients receiving both glucocorticoids and bisphosphonates
  Interventions: Drug: alendronate

INTERVENTIONS:
Drug: alendronate — 70 mg of alendronate orally per week for at least three months in patients receiving at least 10 mg/day or oral prednisone for at least three months
  Other Names: Fosamax; Prednisone
  Groups: glucocorticoids and bisphosphonates

SUMMARY:
The purpose of this study is to determine the difference in response to bisphosphonate therapy in patients receiving excess glucocorticoids compared to patients with postmenopausal or male osteoporosis. Bisphosphonates are approved by the FDA for the treatment of postmenopausal women and osteoporotic men who are at high risk of fracture and in men and women with excess glucocorticoid administration.

DETAILED DESCRIPTION:
Aminobisphosphonates are extensively used to prevent fractures in patients with osteoporosis (1-6). Treatment with these drugs leads to decreases in bone resorption and biochemical markers of bone turnover and progressive increases in bone mineral density (BMD). The increase in BMD in response to bisphosphonate therapy in glucocorticoid-treated patients is, however, less than half that measured in women and men with osteoporosis unrelated to glucocorticoid drugs even though the patients with osteoporosis are usually older. The goal of this objective is to determine the contribution of increased osteoclast survival to the diminished response to bisphosphonate therapy in patients receiving excess glucocorticoids compared to patients with osteoporosis.

1. Liberman U, Weiss SR, Broll J, et al. Effect of oral alendronate on bone mineral density and the incidence of fractures in postmenopausal osteoporosis. N Engl J Med 1995;333:1437-1443.
2. Bone HG, Downs RW, Tucci JR, et al. Dose-response relationships for alendronate treatment in osteoporotic elderly women. J Clin Endocrinol Metab 1997;82:265-274.
3. McClung M, Clemmesen B, Daifotis A, et al. Alendronate prevents postmenopausal bone loss in women without osteoporosis. Ann Intern Med 1998;128:253-261.
4. Recker RR, Weinstein RS, Chestnut CH III, et al. Histomorphometric evaluation of daily and intermittent oral ibandronate in women with postmenopausal osteoporosis: results from the BONE study. Osteoporosis Int 2004;15:231-237.
5. Saag KG, Emkey R, Schnitzer TJ, et al. Alendronate for the prevention and treatment of glucocorticoid-induced osteoporosis. Glucocorticoid-Induced Osteoporosis Intervention Study Group. N Engl J Med 1998;339:292-299.
6. Orwoll E, Ettinger M, Weiss S, et al. Alendronate for the treatment of osteoporosis in men. N Engl J Med 2000;343:604-610.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or greater
2. agree to at least one bone biopsy
3. agree to BMD, blood and urine tests
4. receiving at least 10 mg/day of prednisone for at least three months
5. either be a candidate for alendronate or be taking alendronate (70 mg/week for at least three months)

Exclusion Criteria:

1. any metabolic bone disorder such as Paget's disease, renal osteodystrophy, parathyroid disease or osteomalacia
2. obesity enough to make a biopsy difficult
3. concurrent use of any tetracycline
4. hypercalcemia
5. kidney stones in the last two years
6. home O2
7. gastric surgery, stapling or bypass
8. inflammatory bowel disease
9. untreated thyroid disease
10. organ transplants
11. malabsorption
12. anticoagulation
13. current infection
14. serious illness
15. allergy to Demerol, Valium, iodine, tetracycline, tape
16. use of anticonvulsant drugs, heparin, Forteo, calcitonin or high-dose fluoride within the past six months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults receiving aminobisphosphonate therapy to prevent osteoporosis from glucocorticoids, postmenopausal bone loss or osteoporosis in males
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2004-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jimmie L Valentine, Study Chair — IRB at UAMS
Locations (1):
- University of Arkansas hospitals and clinics and the Central Arkansas Veterans Healthcare System, Little Rock, Arkansas, United States